CLINICAL TRIAL: NCT04939870
Title: Assessment of Protein Modification in Chronic Kidney Disease - Selected Clinical and Biochemical Aspects
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dorota Formanowicz, MD.Ph.D. Associate Professor, Poznan University of Medical Sciences
Other Study IDs: PoznanUMS_DF_1
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Dialysis; Complications
Keywords: oxidative stress, proteins, chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PREDIALYSIS GROUP: (n = 48) - patients in the pre-dialysis period (stage G3b-G4 CKD) with moderate or severe decrease in eGFR (eGFR 44-29 ml / min / 1.73 m2),
  Interventions: Diagnostic Test: Biochemical parameters evaluation
- END-STAGE RENAL DISEASE GROUP: patients with ESRD (n=78) - (eGFR <15 ml/min /1.73 m2) undergoing renal replacement therapy. Depending on the method of renal replacement therapy used, two subgroups are distinguished: PD subgroup (n=35) including patients treated by peritoneal dialysis. In this subgroup, initially, due to the treatment technique, two groups were separated, a group (n=15) treated with the automatic peritoneal dialysis (APD) technique, and a group of patients (n = 20) using the technique of continuous cycling peritoneal dialysis (CCPD), HD subgroup (n = 43) including patients treated with repeated hemodialysis. Hemodialysis procedures were performed in each patient three times a week, via an arteriovenous fistula from own or artificial vessels. The duration of hemodialysis was at least 10 hours/week using standard bicarbonate dialysis fluids and polysulfone low-flux dialyzers. The blood flow during hemodialysis was 200-350 ml/min, with an average dialysis fluid flow of 500 ml/min.
  Interventions: Diagnostic Test: Biochemical parameters evaluation
- CARDIOLOGY GROUP: • CARD group (n = 37) - patients with at least one history of cardiovascular events, admitted to hospital for elective angiography, without any signs of impaired kidney function. The studies in this group were to show the changes that occur as a result of diseases of the cardiovascular system and the functioning of the kidneys.
  Interventions: Diagnostic Test: Biochemical parameters evaluation
- HEALTHY VOLUNTEERS: Healthy volunteers, (n = 32) - it was composed of healthy people, with no evidence of impairment in renal function and cardiovascular function in the history and at the time of enrollment in the study.
  Interventions: Diagnostic Test: Biochemical parameters evaluation

INTERVENTIONS:
Diagnostic Test: Biochemical parameters evaluation — selected biochemical parameters

SUMMARY:
The studies included the effect of chronic kidney disease advancement on the accumulation of oxidative stress markers in plasma. In patients with end-stage renal disease, the effect of replacement therapy was also assessed. Therefore, the patient with chronic kidney disease was evaluated divided into three groups (chronic kidney disease at stage G3b-G4, peritoneal dialysis, hemodialysis). In addition, changes in the interrelationship between oxidative modifications, carbonyl and nitrogen stress, and the carbamylation resulting from the progression of kidney disease have been taken into account. This issue is related to the assessment of whether the protein modification types differentiate patients depending on the stage of chronic kidney disease and the method of renal replacement therapy. Protein modifications associated with oxidative stress are a part of the complications resulting from chronic kidney diseases, such as malnutrition, chronic inflammation, dyslipidemia, iron disorder, and calcium and phosphate disorders. Also, diseases of atherosclerosis aetiology are much higher frequency in patients with chronic kidney disease than in those with normal kidney function. Therefore, in the studies presented here, particular attention was paid to the effect of oxidative stress on chronic kidney disease complications in the aspect of cardiovascular damage. The specificity of atherosclerosis in patients with chronic kidney disease was evaluated by comparing groups of this type of patients with patients with ischemic heart diseases and normal renal function.

DETAILED DESCRIPTION:
Redox imbalance in the course of CKD results in the intensification of oxidative and carbonyl stress, which leads to the modification of many molecules, including proteins necessary for the proper functioning of the body. The assessment of the accumulation of modified proteins in the plasma is not only an indirect indicator of the severity of redox imbalance in the system, but also allows the analysis of the influence of oxidative stress and its derivatives (glycation, carbonyl stress and carbamylation) on the pathogenesis of CKD. In addition, compounds formed as a result of the action of ROS on proteins may affect the development of long-term consequences of CKD, such as chronic inflammation, dyslipidemia, renal osteodystrophy, iron metabolism disorders and malnutrition. On the other hand, complications in patients with CKD may influence the intensification of oxidative modifications of proteins.

The following goals were set in the study:

1. Assessment of the impact of CKD advancement on the severity of protein modification as a result of oxidative stress.
2. Comparison of the effect of renal replacement therapy on protein modifications.
3. Assessment of the relationship between selected protein modifications in CKD and complications typical of CKD
4. Comparison of selected protein modifications in patients with CKD and patients with at least one history of a cardiovascular event.

ELIGIBILITY:
The following criteria of qualifying for the study were adopted for all respondents:

* 18 years of age or older,
* written consent to participate in the study,
* no smoking for at least 10 years in the history of
* no alcohol abuse for at least 10 years in a medical history,
* lack of diabetes and impaired fasting glucose and/or impaired glucose tolerance,
* no active inflammatory process,
* no neoplastic disease or a neoplastic disease whose treatment was stopped at least 10 years ago,
* no history of immunosuppressive treatment,
* stable liver function (not more than two times increased activity of transaminases), HBs antigen and anti-HCV negative antibodies,
* anti-HIV negative antibodies.

In addition, for CKD patients, the following additional inclusion conditions were applied:

* no additional comorbidities that do not result directly or indirectly from CKD,
* no acute cardiovascular complications, ie acute heart failure, hypertensive crisis, acute coronary syndrome, at the time of study entry.

At the same time, depending on the technique of renal replacement therapy used, additional inclusion criteria were established for each of the subgroups:

in group HD:

* a minimum of 6 months of treatment with repeated hemodialysis, 3 times a week, for a minimum of 10 hours a week,
* arteriovenous fistula as a vascular access for hemodialysis,
* Estimated dialysis adequacy ratio (eKt / V) of at least 1.2. in the PD group:
* treatment duration UP to a minimum of 6 months,
* Kt / V ≥1.8 l / week / 1.73 m2.

For CARD patients, additional conditions include:

* no obvious evidence of renal impairment in the history and at the time of study entry, renal function assessed on the basis of eGFR and urine albumin/creatinine ratio,
* history of angina,
* documented history of at least one acute coronary syndrome,
* admission to the Department of Intensive Care of Cardiology and Internal Diseases in order to perform a planned coronary angiography,
* on the day of admission to the study without signs of acute coronary syndrome,
* no additional comorbidities, ie those that do not result directly or indirectly from coronary heart disease.

In turn, for the HV group, additional conditions include:

* no obvious evidence of renal impairment in the history and at the time of study entry, renal function assessed on the basis of eGFR and urine albumin/creatinine ratio,
* no obvious signs of cardiovascular impairment in the history and at the time of study entry, estimated on the basis of normal blood pressure (<140/90 mmHg), no abnormalities in the medical history and physical examination,
* not taking any medications on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study involved 195 people, including 126 patients with diagnosed CKD, under the care of the Nephrology Outpatient Clinic, Peritoneal Dialysis Clinic or the Dialysis Center at the Clinical Hospital. H. Święcicki in Poznań (group from CKD) and 69 people who constituted the control group. Recruitment to the study lasted one year. In the group of patients with CKD, depending on the degree of renal impairment and the type of renal replacement therapy, according to the criteria of diagnosis and classification of CKD according to KDIGO 2012, several subgroups were created. The allocation to groups was based on the GFR, calculated by the recommendations of KDIGO 2012
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters assessed in all groups part 1 | 4 years
  The number of laboratory parameters were determined in all groups:
  * blood count: HGB [g/dl], RBC [10*12/l], HCT [l/l], WBC [10*9/l], PLT [10*9/l]
  * iron metabolism parameters: Fe, UIBC,TIBC [µg/dl], ferritin [ng/ml]
  * glucose [mg/dl]
  * parameters of lipid metabolism [mg/dl] T-C, LDL-C, HDL-C, TG
  * parameters of hepatic metabolism [U/l]: activity of alanine transaminase, aspartate transaminase, alkaline phosphatase
  * creatinine [mg/dl], uric acid [mg/dl], urea [mg/dl],
  * creatinine will be combined with sex [female/male] and age [years] to report eGFR [ml/min/1,73m*2] calculated on the basis on MDRD formula
  * albumin [g/dl] and total protein [g/dl]
  * Na [mmol/l], K [mmol/l]
  * parameters of calcium and phosphate metabolism: total calcium [mg/dl], ionised calcium [mg/dl], phosphates [mg/dl], PTH [pg/ml], FGF-23 [pg/ml], klotho [ng/ml]
  * selected parameters of inflammation: concentration of highly sensitive C-reactive protein (hsCRP) [mg/l]
Biochemical parameters assessed in all groups part 2 - selected parameters of oxidative stress | 4 years
  CML [µg/mg protein], CEL [µg/mg protein], MG [µg/mg protein], AGE [µg/mg protein], RAGE [µg/mg protein] 3-NT [µmol/mg protein], AOPP [µmol/mg protein], carbonyl protein groups [nmol/mg protein], carbamyl protein groups [µg/mg protein]
Demographic data | 4 years
  age [years], sex [number of female and male [n]] were recorded in all groups

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Formanowicz, MD,PhD,Prof, Principal Investigator — Poznan University of Mediccal Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No